CLINICAL TRIAL: NCT01693250
Title: Phase 1 Study of Fitbit and Apps on Healthy Weight Management in Obese Teens in Primary Care Clinics
Brief Title: iStart Smart for Teens for Healthy Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TEENS-2012
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Overweight; Obese
Keywords: technology; healthy weight management; primary care setting
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A randomized control study design with an active control group was used.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Primary care providers and outcome assessors were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fitbit ultra (Experimental): Adolescents in the intervention group will receive a Fitbit Ultra and will download an app to their smartphone. Participants will be asked to wear the Fitbit device and use the app every day for three months.
  Interventions: Behavioral: fitbit Ultra
- Pedometer (Active Comparator): After completion of the baseline assessments, adolescents in the control group will be given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
  Interventions: Behavioral: Pedometer

INTERVENTIONS:
Behavioral: fitbit Ultra — Participants will be asked to wear the Fitbit device and use the app every day for three months. The app functions will include tracking of PA and dietary intake progress, setting individualized and realistic goals, monitoring progress related to reaching the goals, providing tips of everyday activities, and having interactive games related to PA and healthy diet.
  Other Names: Fitbit Ultra and associated apps
  Arms: fitbit ultra
Behavioral: Pedometer — adolescents in the control group will be given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
  Other Names: Omron HJ-105 pedometer
  Arms: Pedometer

SUMMARY:
The emerging epidemic of type 2 diabetes mellitus (T2DM) in children is coupled with the increased prevalence of childhood obesity in the last two decades. Obesity during the adolescent years is associated with many adverse health consequences, including T2DM, hyperlipidemia, and psychosocial problems. The first step toward effective obesity management and T2DM prevention is monitoring of physical activity (PA) and dietary intake. With the rapid expansion of cellular networks, and advancements in smartphone technologies, it is now possible to monitor PA and dietary intake and at the same time to transmit data digitally to their primary care providers (PCP). The proposed pilot study will include the collaboration among UCSF, North East Medical Services (NEMS), mHealth teams, and overweight and/or obese adolescents. The study will adapt and implement smartphone-based technologies and integrate these technologies with the Electronic Health Record (EHR) to increase PA and dietary intake. Two specific aims of this proposed study include: (1) adapt fitbit Ultra applications for the smartphone-based technologies and EHR and (2) and assess the feasibility and estimate the effect for patient outcomes (self-efficacy, physical activity, dietary intake, BMI, and lipid profile), at 3 months post intervention between the intervention and control groups. The smartphone app for the intervention group will allow the teens to graphically compare daily PA and dietary intake with the goal, participate in a reward program where they can collect virtual points for achieving the goal, and play interactive games related to PA and diet. A total of 40 overweight and/or obese adolescents at NEMS will be recruited and randomized to the feasibility study (Aim 2).

DETAILED DESCRIPTION:
Using evidence to inform the design of clinical practice is a foundational principle of modern health care practice. In the present pilot study, using evidence from research on technology in clinical practice facilitated development of a hybrid intervention that combined lifestyle modification with routine clinical care. Chief among the benefits of this hybrid smartphone technology-based intervention (STB) was the potential to improve health outcomes and reduce obesity in overweight and obese adolescents. The purposes of this study were to (1) measure effects of an innovative smartphone-technology-based (STB) intervention for overweight and obese adolescents and to (2) examine the intervention's feasibility for use in primary care clinics.The STB intervention had 3 components: use of Fitbit Flex, participation in the online educational program, and receipt of bi-weekly text message during the maintenance phase. A randomized control study design was utilized. Data regard to anthropometrics (BMI and waist-hip ratio), blood pressure, levels of physical and sedentary activity, diet, and self-efficacy regarding physical activity and diet were collected at baseline, 3 month and 6 months after the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* between 13-18 years old
* have a BMI at ≥ 85th percentile, based on CDC growth chart
* own a smartphone;
* have access to a computer with internet access
* be able to read and speak English.

Exclusion Criteria:

* have acute or life-threatening disease
* not be able to engage in activities of daily living

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyu-Lin Chen, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF School of Nursing, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karnik S, Kanekar A. Childhood obesity: a global public health crisis. Int J Prev Med. 2012 Jan;3(1):1-7. PMID 22506094
- [Background] Wang LY, Chyen D, Lee S, Lowry R. The association between body mass index in adolescence and obesity in adulthood. J Adolesc Health. 2008 May;42(5):512-8. doi: 10.1016/j.jadohealth.2007.10.010. Epub 2008 Jan 31. PMID 18407047
- [Background] Chen JL, Wilkosz ME. Efficacy of technology-based interventions for obesity prevention in adolescents: a systematic review. Adolesc Health Med Ther. 2014 Aug 7;5:159-70. doi: 10.2147/AHMT.S39969. eCollection 2014. PMID 25177158
- [Background] Chen JL, Weiss S, Heyman MB, Cooper B, Lustig RH. The efficacy of the web-based childhood obesity prevention program in Chinese American adolescents (Web ABC study). J Adolesc Health. 2011 Aug;49(2):148-54. doi: 10.1016/j.jadohealth.2010.11.243. Epub 2011 Mar 12. PMID 21783046
- [Background] Delamater AM, Pulgaron ER, Rarback S, Hernandez J, Carrillo A, Christiansen S, Severson HH. Web-based family intervention for overweight children: a pilot study. Child Obes. 2013 Feb;9(1):57-63. doi: 10.1089/chi.2011.0126. Epub 2013 Jan 11. PMID 23308372
- [Background] Sim LA, Lebow J, Wang Z, Koball A, Murad MH. Brief Primary Care Obesity Interventions: A Meta-analysis. Pediatrics. 2016 Oct;138(4):e20160149. doi: 10.1542/peds.2016-0149. Epub 2016 Sep 12. PMID 27621413
- [Background] Al-Khudairy L, Loveman E, Colquitt JL, Mead E, Johnson RE, Fraser H, Olajide J, Murphy M, Velho RM, O'Malley C, Azevedo LB, Ells LJ, Metzendorf MI, Rees K. Diet, physical activity and behavioural interventions for the treatment of overweight or obese adolescents aged 12 to 17 years. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012691. doi: 10.1002/14651858.CD012691. PMID 28639320
- [Result] Chen JL, Guedes CM, Lung AE. Smartphone-based Healthy Weight Management Intervention for Chinese American Adolescents: Short-term Efficacy and Factors Associated With Decreased Weight. J Adolesc Health. 2019 Apr;64(4):443-449. doi: 10.1016/j.jadohealth.2018.08.022. Epub 2018 Nov 6. PMID 30409751
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Chen JL, Guedes CM, Cooper BA, Lung AE. Short-Term Efficacy of an Innovative Mobile Phone Technology-Based Intervention for Weight Management for Overweight and Obese Adolescents: Pilot Study. Interact J Med Res. 2017 Aug 2;6(2):e12. doi: 10.2196/ijmr.7860. PMID 28768612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trained research assistant worked with primary care providers at two large community clinics whose patient populations were predominantly Chinese American in northern California. A study invitation letter was posted in the clinics. Pediatricians at the clinics were also given a study invitation letter to give to potential participants.
Pre-assignment Details: An explanation of why potential participants were excluded from the study before assignment to groups was given them.
Groups:
- Fitbit Ultra: A total of 23 adolescents in the intervention group received a Fitbit Ultra and will download an app to their smartphone. Participants will be asked to wear the Fitbit device and use the app every day for three months.
  fitbit Ultra: Participants were asked to wear the Fitbit device and use the app every day for three months. The app functions will include tracking of PA and dietary intake progress, setting individualized and realistic goals, monitoring progress related to reaching the goals, providing tips of everyday activities, and having interactive games related to PA and healthy diet.
- Pedometer: A total of 17 adolescent included in the control group. After completion of the baseline assessments, adolescents in the control group were given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
  Pedometer: adolescents in the control group were given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
Period: Overall Study
Arm/Group | Fitbit Ultra | Pedometer
Started | 23 (3 months post baseline assessment) | 17 (three month post baseline assessment)
Completed | 21 (21 teens completed 6 months post baseline assessment) | 15 (15 teens completed 6 months post baseline assessment)
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: 23 participants were assigned to the fitbit ultra group and 17 were assigned to Pedometer group
Groups:
- Total: Total of all reporting groups
Arm/Group | Fitbit Ultra | Pedometer | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 17 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.66) | 14.8 (1.69) | 14.9 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: Participants' BMI was determined by dividing body mass (weight) by height squared (kg/m2). Adolescents' weight and height were measured while the adolescents wore light-weight clothes and no shoes. For BMI, adequate sensitivity and specificity has been reported in children and adolescents, with sensitivity ranging from 29% to 88% and specificity ranging from 94% to 100%.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Fitbit Ultra: Participants in the intervention group received a Fitbit Ultra and will download an app to their smartphone. Participants will be asked to wear the Fitbit device and use the app every day for three months.
  fitbit Ultra: Participants were asked to wear the Fitbit device and use the app every day for three months. The app functions will include tracking of PA and dietary intake progress, setting individualized and realistic goals, monitoring progress related to reaching the goals, providing tips of everyday activities, and having interactive games related to PA and healthy diet.
- Pedometer: After completion of the baseline assessments, adolescents in the control group were given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
  Pedometer: adolescents in the control group were given an Omron HJ-105 pedometer and a food diary and be asked to use them for three months.
Arm/Group | Fitbit Ultra | Pedometer
Number analyzed (Participants) | 23 | 17
kg/m^2
  baseline data | 27.37 (3.26) | 28.35 (4.36)
  6 months data | 26.93 (3.42) | 29.18 (3.88)
Statistical Analysis 1: Comparison: Fitbit Ultra vs Pedometer; This is a feasibility and pilot study. We acknowledge that our sample size will not have adequate power to detect any statistically significant outcomes. We chose a sample size that would be large enough to assess feasibility and effect size and to accommodate recruitment within the study time and budget of this application. We hope to be able to estimate the effect size of the intervention; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 1.68, Standard Deviation .5

2. Other Pre Specified Outcome: Diastolic Blood Pressure
Description: Systolic blood pressure and diastolic blood pressure were measured by using a mercury sphygmomanometer with specific cuff size appropriate for adolescents (Baumanometer, W. A. Baum Co., Copiague, New York). After participants sat for 10 minutes, blood pressure was measured twice in the adolescent's right arm; blood pressures were measured to the nearest 2 mmHg. Average score of two measures was used.
Time Frame: baseline and 6 months
Population: Adolescents who are overweight or obese were invited to participate in this study,
Measure: Mean (Standard Deviation); unit: mmhg
Arm/Group | Fitbit Ultra | Pedometer
Number analyzed (Participants) | 23 | 17
mmhg
  baseline | 72.74 (8.07) | 69.94 (11.25)
  6 month | 70.15 (7.53) | 72.14 (8.71)
Statistical Analysis 1: Comparison: Fitbit Ultra vs Pedometer; We hypothesized the intervention group will have significant reduction of systematic blood pressure compared to the control group at 6 month follow up; Test type: Superiority; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = 2.66

ADVERSE EVENTS:
Time Frame: The study period is 6 months, therefore, adverse event data were collected over 6 months.
Description: Any adverse event happened during the study period will be reported to UCSF Institutional Review Board. The IRB will review the adverse event report and determine if a) the risk-benefit ratio continues to be acceptable, b) the research protocol and informed consent document accurately and completely present risk information, c) current subjects should be advised of newly identified risks and d) the event meets the definition of an Unanticipated Problem involving risk to participants or others.
Arm/Group | Fitbit Ultra | Pedometer
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/17
Other Adverse Events (participants affected / at risk) | 0/23 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No